CLINICAL TRIAL: NCT03436381
Title: Can a Higher Body Mass Index and a Positive Stop Bang or Epworth Sleepiness Scale Questionnaire Predict Cardiorespiratory Adverse Events During Endoscopy: A Prospective Cohort Study
Brief Title: Can Sleep Apnea Screening Questionnaire Predict Adverse Events in Endoscopic Studies
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Fernando Castro, M.D., The Cleveland Clinic
Other Study IDs: FLA 17-104
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2019-12

CONDITIONS: Sleep Apnea; Adverse Event
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Overweight and obese patients: Patient undergoing elective upper endoscopy or colonoscopy, body mass index equal or greater than 25 kg/m2.
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — We will provide two sleep apnea screening questionnaire, Stop-bang questionnaire and Epworth sleepiness scale

SUMMARY:
Investigators hypothesize that the obese population (BMI ≥30 kg/m2) who might be at higher risk for obstructive sleep apnea (OSA), carries a higher risk of endoscopy associated adverse events. The primary aim of our study is to determine predictors of endoscopy associated adverse events (airway maneuvers and sedation related complications) in the obese population including the use of the STOP-BANG questionnaire (SBQ) and Epworth Sleepiness Scale (ESS). A secondary aim is to determine the impact of referral to sleep medicine clinic and home sleep test ordered from the gastroenterologist if patient was found to be high risk for OSA by the use of validated questionnaires such as SBQ and ESS.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a chronic condition characterized by episodes of apnea and hypoxemia caused by upper airway collapse. These episodes lead to symptoms such as daytime fatigue and sleepiness in addition to multiple effects on health including hypertension, stroke, cardiovascular disease and diabetes. Obesity, defined by the World Health Organization and the United States National Institute of Health as a body mass index (BMI) ≥30 kg/m2 is a major risk factor for OSA and along with the obesity epidemic, the prevalence of OSA has been increasing and is estimated to be around 3-7% in the United States. In 2017 The American Gastroenterological Association release the Practice guide on Obesity and Weight management, Education and Resources (POWER) that provides guidance on obesity management. This is in recognition that gastroenterologists are at the frontline of managing patients with multiple obesity related conditions such as non-alcoholic fatty liver disease, non-alcoholic steatohepatitis, gastroesophageal reflux, Barrett's esophagus, and colon cancer. In the midst of these guidelines, recognition of extra gastrointestinal obesity related conditions such as OSA remains an important task as this can have important long-term health consequences.

There are different tools modalities to screen for OSA such as STOP-BANG questionnaire (SBQ) and the Epworth Sleepiness scale (ESS). The SBQ was originally developed to screen patients in the pre-operative setting as this population may be at higher risk for post-operative complications, however this tool has been validated by multiple studies to identify patients that may be at high risk for OSA. A systematic review and meta-analysis on the performance of SBQ in different populations showed a sensitivity of 90%, 94% and 96% to detect any OSA (Apnea-Hypopnea Index (AHI) ≥ 5), moderate-to-severe OSA (AHI ≥15), and severe OSA (AHI ≥30) respectively. The ESS is a simple and validated questionnaire for assessing excessive daytime sleepiness in the context of sleep disorders and has been suggested as a tool to identifying patient with OSA. Studies comparing ESS with SBQ showed that although SBQ identify more patient with OSA, the ESS has a higher specificity which is potentially of use in conjunction with another higher sensitivity modality such as SBQ may improve the diagnostic accuracy other screening modalities. Although the sensitivity of Berlin, STOP and STOP-Bang questionnaires was generally high, the low specificity of these questionnaires results in increased false positives and failure of exclusion of individuals at low risk.

The high sensitivity of SBQ, high specifity of ESS and ease in performing these questionnaire makes it an ideal tool to screen patients for OSA in the endoscopy unit. Given the potential cardiorespiratory decompensations in patients with OSA, multiple studies have used this questionnaire to determine factors associated with airway maneuvers (AM) and sedation related complications (SRC). In one study of patients undergoing advanced endoscopic procedures a SBQ score ≥3 (SBQ+) was associated with increased risk of hypoxemia and the use of AM. These patients also had a mean BMI of 31.4 kg/m2 which is defined as obesity class I. A similar study on patients undergoing elective EGD and colonoscopy found no correlation between SBQ+ patients and SRC or AM, however it should be noted that the mean BMI in this SBQ+ population was 28.3 kg/m2 which does not meet criteria for obesity. Although not statistically significant there was a trend towards a higher use of AM in the higher BMI group (p=0.066). In addition the combined analysis of adverse events for EGD and colonoscopies together can be problematic since only about half of the patients on the study (n=120) underwent EGD which has a higher risk of transient hypoxemia than colonoscopy, because of the potential of direct impingement of the airway, laryngeal irritation or micro aspiration during esophageal intubation17. Also the use of propofol was not standardized and other methods of sedation were used such as benzodiazepine and opioids.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective upper endoscopy or colonoscopy
2. Body mass index equal or greater than 25 kg/m2

Exclusion Criteria:

1. Patients <18 years of age
2. pregnant women
3. lung disease requiring oxygen
4. oxygen saturation less or equal to 90% at the beginning of endoscopy
5. BMI <25
6. ASA ≥4
7. Inability to obtain consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient presenting to endoscopy unit for routine esophagogastrodudenoscopy, colonoscopy or both who have a BMI equal or greater than 25 kg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Predictors of endoscopy associated adverse events | 2/9/2018 - 2/18/2019
  Determine predictors of endoscopy associated adverse events (airway maneuvers and sedation related complications) in the obese population including the use of the STOP-BANG questionnaires and Epworth sleepiness scale

SECONDARY OUTCOMES:
Impact of referral to sleep medicine clinic and home sleep test | 2/9/2018 - 2/18/2019
  Determine the impact of referral to sleep medicine clinic and home sleep test ordered from the gastroenterologist if patient were found to be high risk for OSA by the use of validated questionnaires such as STOP-BANG questionnaire and Epworth sleepiness questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Castro, M.D, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided